CLINICAL TRIAL: NCT05909059
Title: Lymphodepleting Chemotherapy With Fludarabine and Cyclophosphamide Prior to Infusion of CAR T Cell Therapy in Patients With Moderate-Severe Renal Dysfunction
Brief Title: CAR T-cell Therapy in Patients With Renal Dysfunction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Blood and Marrow Transplant Group of Georgia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1375
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Non-hodgkin Lymphoma,B Cell; Multiple Myeloma; Acute Lymphoblastic Leukemia, Adult
MeSH Terms: conditions — Multiple Myeloma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Moderate Renal Dysfunction (Experimental): Moderate renal dysfunction will receive a 20% dose reduction of fludarabine and no dose reduction for cyclophosphamide.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide
- Severe Renal Dysfunction (Experimental): Several renal dysfunction will receive a 40% dose reduction of fludarabine and no dose reduction for cyclophosphamide.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide
- Dialysis Participants (Experimental): Participants on dialysis will receive a 50% dose reduction of fludarabine and a 25% dose reduction of cyclophosphamide.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Fludarabine — Received IV on Days -5 to -3 before CAR T cell therapy
Drug: Cyclophosphamide — Received IV on Days -5 to -3 before CAR T cell therapy

SUMMARY:
This is a prospective, descriptive study designed to assess the feasibility of administering CAR T therapy among patients with moderate to severe renal impairment using dose adjusted lymphodepleting chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Receiving lymphodepleting chemotherapy prior to commercial CAR-T administration for multiple myeloma, leukemia, or lymphoma
* Adequate bone marrow function to receive lymphodepleting chemotherapy
* Renal function </= 60mL/min/1.73m2
* ECOG 0-2

Exclusion Criteria:

* Relative CNS disorders
* Active uncontrolled infection or any other concurrent disease or medical condition that was deemed to interfere with the conduct of the study as judged by the investigator
* Use of therapeutic dose systemic corticosteroids (defined as >20mg/day prednisone or equivalent) within 72 hours of CAR-T administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of CRS | 90 days
  Collection of maximum grade of CRS (based on CTCAE v5) and when this event occurs post CAR T cell therapy infusion
Occurrence of ICANS | 90 days
  Collection of maximum grade of ICANs (based on CTCAE v5) and when this event occurs after CAR T cell therapy infusion
Occurrence of Cytopenias | 90 days
  Collection of grade 3 or higher (based on CTCAE v5) cytopenias not resolved by Day 30 post CAR T cell infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Caitlin Guzowski, Atlanta, Georgia, United States